CLINICAL TRIAL: NCT04387396
Title: Investigation of the Effects of Physiotherapy on Pain, Physical Function and Quality of Life in Patients With PRP Applied Knee Osteoarthritis
Brief Title: Investigation of the Effects of Physiotherapy in Patients With Platelet Rich Plasma (PRP) Applied Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Sibel Bozgeyik, PT, PhD(c), Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KA-180151
Record Dates: First submitted 2019-10-24; First posted 2020-05-13 (Actual); Last update posted 2021-02-16 (Actual); Status verified 2021-02

CONDITIONS: Knee Osteoarthritis
Keywords: Knee Osteoarthritis; Platelet rich plasma; Exercise
MeSH Terms: conditions — Osteoarthritis, Knee; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physiotherapy (Experimental): Exercise intervention will be applied to this arm.
  Interventions: Other: Exercise
- Control (No Intervention): No intervention will be made to this arm, only evaluations will be made.

INTERVENTIONS:
Other: Exercise — Exercise specific to knee osteoarthritis.
  Arms: Physiotherapy

SUMMARY:
This study evaluates effects of PRP and physiotherapy on pain, physical function and quality of life in patients with knee osteoarthritis.

DETAILED DESCRIPTION:
PRP has been reported to have a low to moderate level of evidence in patients with knee osteoarthritis (OA) in reducing pain and improving function. Similarly, in individuals with knee osteoarthritis, exercise has been reported to be effective in reducing the pain and improving physical function of the knee OA patient in the short term, and may be even more effective with individual exercise programs. However, there is no study examining the effect of PRP and exercise together. PRP and exercise can be more effective together. The aim of our study was to investigate the effects of physiotherapy on pain, physical function and quality of life in patients with knee OA who underwent PRP injection.

ELIGIBILITY:
Inclusion Criteria:

* Grade 2-3 according to Kellgren Lawrence osteoarthritis classification,
* Patients with knee osteoarthritis who underwent PRP injection at least three days ago,
* Being volunteer

Exclusion Criteria:

* Any intra-articular application and / or physiotherapy and rehabilitation in the last 6 months,
* Have any other orthopedic problems involving the lower extremities
* Having cognitive problems,
* Having additional neurological, rheumatologic and / or oncological problems

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 26 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-12-29 (Actual); Study Completion 2020-12-29 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Pain Level at Six Week | At baseline, six week
  Pain change will be measured throughout Study and Follow-up with Visual Analog Scale. This scale is a 100 millimeter line drawn horizontally on an A4 sheet of paper. The left end of the line shows "no pain at all", the right end shows "my pain is as bad as it could be", while the remaining part shows the intermediate values. So minimum score was 0, and maximum score was 100. The patient is asked to mark the severity of the pain on the chart. Validity and reliability were made. The minimal clinical significance difference in chronic low back pain was 20 millimeters.

CONTACTS AND LOCATIONS:
Overall Officials: Feza Korkusuz, Prof., Principal Investigator — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Samanpazari, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Recommendations for the medical management of osteoarthritis of the hip and knee: 2000 update. American College of Rheumatology Subcommittee on Osteoarthritis Guidelines. Arthritis Rheum. 2000 Sep;43(9):1905-15. doi: 10.1002/1529-0131(200009)43:93.0.CO;2-P. No abstract available. PMID 11014340
- [Background] MILLER JH, WHITE J, NORTON TH. The value of intra-articular injections in osteoarthritis of the knee. J Bone Joint Surg Br. 1958 Nov;40-B(4):636-43. doi: 10.1302/0301-620X.40B4.636. No abstract available. PMID 13610976
- [Background] Bennell KL, Hunt MA, Wrigley TV, Lim BW, Hinman RS. Role of muscle in the genesis and management of knee osteoarthritis. Rheum Dis Clin North Am. 2008 Aug;34(3):731-54. doi: 10.1016/j.rdc.2008.05.005. PMID 18687280
- [Background] Laudy AB, Bakker EW, Rekers M, Moen MH. Efficacy of platelet-rich plasma injections in osteoarthritis of the knee: a systematic review and meta-analysis. Br J Sports Med. 2015 May;49(10):657-72. doi: 10.1136/bjsports-2014-094036. Epub 2014 Nov 21. PMID 25416198
- [Background] Chang TF, Liou TH, Chen CH, Huang YC, Chang KH. Effects of elastic-band exercise on lower-extremity function among female patients with osteoarthritis of the knee. Disabil Rehabil. 2012;34(20):1727-35. doi: 10.3109/09638288.2012.660598. Epub 2012 Mar 8. PMID 22397710

DOCUMENTS (1):
  • Statistical Analysis Plan (2019-06-24): https://cdn.clinicaltrials.gov/large-docs/96/NCT04387396/SAP_000.pdf